CLINICAL TRIAL: NCT05668494
Title: Immediate Loading With Provisional Prosthetic Restoration by Means of One Abutment at One Time and Temporary Abutment in the Posterior Mandible Without Bone Augmentation
Brief Title: Immediate Loading With Provisional Prosthetic Restoration by Means of One Abutment at One Time and Temporary Abutment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Ana Todorovic, Principal Investigator, University of Belgrade
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: One abutment one time study
Record Dates: First submitted 2022-12-05; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Bone Loss in Jaw

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immediate loading (Other): Immediate loading of implants by means of one definitive abutment on one side and temporary abutment on the other side of the posterior mandible restored by provisional crown-split mouth design
  Interventions: Other: immediate loading of implants

INTERVENTIONS:
Other: immediate loading of implants — This is a randomized control clinical trial including 24 implants, immediately loaded with definitive abutment protocol and 24 implants immediately loaded with with temporary abutment protocol

SUMMARY:
This will be a prospective, randomized, controlled, single center clinical trial with

1 year enrollment period, surgical and prosthetic rehabilitation with 1-year post-loading follow-up. A total of 2.0 years of study duration The primary objective is to compare peri-implant hard and soft tissue changes between single implants placed in the posterior mandible and immediately loaded either with definitive (one-time) or provisional abutment.

DETAILED DESCRIPTION:
Hard tissue contour changes will be assessed using standardized two-dimensional intra-oral radiographs and partial small field of view three-dimensional cone beam CT scans. Soft tissue contour changes will be assessed using superimposition of dental digital models. Inflammatory soft tissue reactions will be evaluated by measurement of respective cytokines' levels.A quantitative evaluation of total bacteria amount of the peri-implant samples.

Secondary objectives of this study will be to estimate total bacterial amount (quantitative real-time polymerase chain reaction - qRT-PCR).

Bleeding on probing (BoP), full mouth oral hygiene index, periodontal pocket depth (PPD) and keratinized tissue width will also be evaluated.

Indication: Patients with need of at least two implants (one per side) in the premolar or molar region in the mandible, bilaterally.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 25 years
* In need of a one or two implants.
* Healed site (healed site defined by restored gingiva, free of inflammation and scar tissue , with a keratinized band of 3mm from crest to muco-gingival junction, and sufficient osseous architecture to receive an implant with a minimal diameter of 3.5 mm).
* Mandible second premolar or molar region.
* At least one neighboring tooth to be present.
* Absence of visible active periapical or periodontal inflammation.
* Adequate oral hygiene: PI< 20%, BoP< 20%.
* Sufficient occlusal units mesial or distal and antagonizing, including the diastema to be restored: 4 occlusal units.

Exclusion Criteria:

* Medical condition that contraindicates surgery: ASA -score ≥ III
* History of radiotherapy in the head and neck region.
* History of Bisphosphonate medication.
* Medium smokers ≥ 10 cigarettes per day.
* Patients unwilling or incapable of understanding and signing the informed consent.
* Active caries.
* Presence of inflammation expressed by PPD >4mm and BoP on adjacent teeth.
* Active periapical radiolucency or root canal treatment performed < 4 months previous to planned implant insertion on a neighboring tooth to future implant.
* Insufficient restorative space.
* Interocclusal plane distance < 20mm at planed implant position.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Periimplant marginal bone loss | 12 months
  Hard tissue changes will be analyzed and followed up at 3, 6 and 12 months by captured intraoral radiographs using a customized radiographic holder. The following landmarks will be measured in order to assess bone remodelling around implants
  * Mesial distance in mm from first bone to implant contact to implant shoulder (vertical line);
  * Distal distance in mm from first bone to implant contact to implant shoulder (vertical line) after implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Ana R Todorovic, DDS,PhD, Principal Investigator — School of Dentistry, University of Belgrade
Locations (1):
- School of Dental Medicine University of Belgrade, Belgrade, Serbia